CLINICAL TRIAL: NCT02304549
Title: Is Absorption of Irrigation Fluid a Problem in Thulium Laser Vaporization of the Prostate? A Prospective Investigation Using the Expired Breath Ethanol Test.
Brief Title: A Prospective Investigation Using the Expired Breath Ethanol Test
Status: Completed | Type: Observational
Sponsor: Daniel Stephan Engeler (Other)
Responsible Party: Sponsor-Investigator, Daniel Stephan Engeler, Dr. med., Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Other Study IDs: CTU 14.012
Record Dates: First submitted 2014-11-17; First posted 2014-12-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Benign Prostatic Hyperplasia (BPH)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with BPH undergoing TUV-P: patients with Benign Prostatic Hyperplasia undergoing TUV-P

SUMMARY:
Benign prostatic hyperplasia (BPH) is a prevalent entity, affecting over 50% of men older than 60 years.In cases with moderate to severe lower urinary tract symptoms (LUTS) monopolar transurethral resection of the prostate (TUR-P) is the standard treatment. Especially in frail patients, conventional TUR-P is associated with relevant and potentially deleterious complications, e.g. TUR syndrome. Using isotonic saline, like in bipolar TUR-P and transurethral laser vaporization (TUV-P), TUR syndrome can be prevented.

The short-term complication rate with the Thulium laser is similar to the rate described after vaporisation with other laser systems18-23 and less than that with TUR-P.

Despite recent publications on the safety and complications with Thulium vaporisation of the prostate, to the investigators knowledge, until now, no prospective trial has directly assessed, whether absorption of irrigation fluid occurs and to what extent in Thulium Laser vaporisation of the prostate.

The investigators therefore aim to investigate if absorption of irrigation fluid occurs during Thulium Laser vaporisation of the prostate by expired breath ethanol test.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is a prevalent entity, affecting over 50% of men older than 60 years.3 The clinical picture of the disease includes lower urinary tract symptoms such as interrupted and weak urinary stream, nocturia, urgency and leaking and even sexual dysfunction in some individuals. Medical therapy is usually the first-line treatment. However, the efficacy of drugs like alpha-blockers is limited, and as disease progresses more invasive treatment options have to be taken into consideration.

In cases with moderate to severe lower urinary tract symptoms (LUTS) monopolar transurethral resection of the prostate (TUR-P) is the standard treatment. Especially in frail patients, conventional TUR-P is associated with relevant and potentially deleterious complications.

The proportion of elderly patients on anticoagulation or antiplatelet therapy with cardial comorbidities increases. Especially major bleeding and transurethral resection syndrome (TUR syndrome) put these high-risk patients at a relevant perioperative risk.

TUR syndrome is caused by absorption of electrolyte-free irrigating fluid (which has to be used in monopolar TUR-P), and consists of symptoms from the circulatory and nervous systems. Mild forms are common and often go undiagnosed, while severe forms of the TUR syndrome are potentially life-threatening.

Using isotonic saline, like in bipolar TUR-P and transurethral laser vaporization (TUV-P), TUR syndrome can be prevented. Moreover, these techniques were thought to completely prevent influx of irrigation fluid into the vascular system due to their excellent coagulation properties.

However, the Zürich study group has demonstrated that in bipolar resection of the prostate and with the Greenlight-Laser, significant intraoperative fluid absorption can occur. The authors emphasized, that care must be taken if using this procedures in patients with significant cardiovascular comorbidities, as large volume influx in patients with significant cardiac comorbidities could result in dangerous complications.

Ethanol monitoring was first used in the late 1980's as an alternative to traditional methods of measuring fluid absorption (i.e. measuring volumetric fluid balance and serum sodium concentration). These techniques, however, are bothersome and must be carried out meticulously to yield a valid figure of absorption. If a tracer amount of ethanol is added to the irrigation fluid, the volume of fluid absorbed can be estimated from the amount of ethanol measured in the patients' exhaled breath.

The expired-breath ethanol technique is an established method of investigating intra operative absorption of irrigation fluid. Ethanol 1% is added to conventional isotonic 0.9% saline for use as intra-operative irrigation. The absorption of irrigation fluid can be estimated by measuring the end-expiratory ethanol concentrations with an alcometer.

During the last years, the Thulium laser has emerged as an alternative to other types of lasers, combining the best features for performing vaporisation techniques: Thulium laser has a wavelength of 2013 nm, and its target chromophore is water. The energy of the Thulium laser has a high tissue absorption rate, producing effective vaporisation with scant depth in the remaining tissue. As the properties of water remain unaltered until it reaches boiling point, the effect of the laser on the tissue remains constant throughout the surgical procedure.

The short-term complication rate with the Thulium laser is similar to the rate described after vaporisation with other laser systems and less than that with TUR-P. Thus, Thulium vaporisation of prostate has established as a standard procedure in many urological departments including ours.

Despite recent publications on the safety and complications with Thulium vaporisation of the prostate, to the investigators knowledge, until now, no prospective trial has directly assessed, whether absorption of irrigation fluid occurs and to what extent in Thulium Laser vaporisation of the prostate.

The investigators therefore aim to investigate if absorption of irrigation fluid occurs during Thulium Laser vaporisation of the prostate by expired breath ethanol test.

ELIGIBILITY:
Inclusion Criteria:

* Men older than 40
* Patient must be a candidate for TUV-P
* Refractory to medical therapy or patient is not willing to consider (further) medical treatment
* Written informed consent

Exclusion Criteria:

* Mild symptoms (IPSS <8)
* Urethral stenosis
* Bladder diverticulum (>100ml)
* Former alcoholic or chronic liver disease
* Alcohol consumption 24h before operation

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with benign prostatic hyperplasia undergoing TUV-P
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Absorption volume of irrigation fluid during the Thulium laser TUV-P | shortly after Thulium laser TUV-P

SECONDARY OUTCOMES:
Duration of surgery | at time of start and of end of surgery
Does absorption of irrigation fluid occur? | at time of surgery
  yes: any detection of alcohol in the expired breath
Assessment of bleeding and relevant intraoperative events (capsular perforation, injury to prostatic sinuses or deep bladder neck incision) by the surgeon | at time of surgery
Amount of laser energy used intraoperatively (kilojoules) | at time of end of surgery
Pre- to postoperative changes in serum biochemical and haematological variables (creatinin, sodium, potassium, chloride), venous pH, haemoglobin | 30 min after intervention
Pre- to postoperative changes in flow and residual urine | 12 weeks after intervention
Total irrigation volume and volume of all administered i.v. fluids | at time of end of surgery
Duration of hospitalization post procedure | participants will be followed for the duration of hospital stay, an expected average of 1 week
Duration of post procedure catheterization | at time of end of catheterization, an expected average of 48 hrs
Pre- to postoperative changes in the IPSS | 12 weeks after intervention
Pre- to postoperative changes in bladder diary | 12 weeks after intervention

OTHER OUTCOMES:
Adverse events categorised according to the NCI-CTAE in grade 1 to 5 | week 12
Grading of complications according to Clavien classification | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Engeler, MD, Study Chair — Cantonal Hospital of St. Gallen
Locations (1):
- Cantonal Hospital St. Gallen, Sankt Gallen, Switzerland

REFERENCES:
- [Background] Mordasini L, Abt D, Mullhaupt G, Engeler DS, Luthi A, Schmid HP, Schwab C. Is absorption of irrigation fluid a problem in Thulium laser vaporization of the prostate? A prospective investigation using the expired breath ethanol test. BMC Urol. 2015 Apr 24;15:35. doi: 10.1186/s12894-015-0029-2. PMID 25903582